CLINICAL TRIAL: NCT02223221
Title: Effects of Preimplantation Genetic Screening for Aneuploidies in Infertile Female Patients With Recurrent Spontaneous Abortion History
Brief Title: Effects of PGS in Infertile Female Patients With RPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JIAI E2014-02
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Infertility, Female; Abortion, Habitual
Keywords: In Vitro Fertilization; Intracytoplasmic Sperm Injections; Infertility, Female; Abortion, Habitual; recurrent pregnancy loss; comprehensive chromosome screening; preimplantation genetic screening; SNP array
MeSH Terms: conditions — Infertility, Female; Abortion, Habitual | interventions — Phosphatidylglycerols

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With PGS (Experimental): IVF/ICSI cycles with PGS. Select embryos by SNP-array based PGS for the number of all chromosomes on day 5, only euploid embryos will be transferred.
  A maximum of 2 embryos will be transferred for each treatment cycle. Up to 3 treatment cycles will be offered.
  Interventions: Procedure: IVF/ICSI; Genetic: PGS
- Without PGS (Active Comparator): IVF/ICSI cycles without PGS. Selection of embryos are based on blastocyst morphology criteria on day 5.
  A maximum of 2 embryos will be transferred for each treatment cycle. Up to 3 treatment cycles will be offered.
  Interventions: Procedure: IVF/ICSI; Other: Without PGS

INTERVENTIONS:
Procedure: IVF/ICSI — In vitro fertilization or intracytoplasmic sperm injection.
Genetic: PGS — Selection of embryos are based on SNP-array-based preimplantation genetic screening for the number of all chromosomes on the 5th day of IVF/ICSI.
  Arms: With PGS
Other: Without PGS — Selection of embryos are based on morphology criteria on the 5th day of IVF/ICSI.
  Arms: Without PGS

SUMMARY:
Recurrent pregnancy loss (RPL) is a multifactorial disorder which affects about 1% of all couples and challenges both patients and clinicians technically and emotionally. IVF clinics see higher prevalence of RPL, since many RPL patients are seeking for assist reproduction treatment with or without other infertile factors. Guidelines for evaluation and treatment of RPL patients include screening for uterine abnormalities, parental chromosomes, autoimmune antibodies and cure gynecological infections, but there are still half of RPL patients remain unexplained.

The documented high incidence of chromosomal errors in first-trimester miscarriages and an increased rate of aneuploidy in patients with RPL has led to the theory that screening embryos before implantation for aneuploidy may decrease the risk of a subsequent loss and serve as a possible treatment. The technology, indications of use, and even terminology for genetic testing of embryos have greatly changed since the first PGD(pre-implantation genetic diagnosis) baby was born in 1990. The current best evidence shows blastocyst biopsy followed by new rapid comprehensive chromosome screening(termed pre-implantation chromosomal screening or comprehensive chromosome screening, PCS or CCS, or the investigators generally termed PGS) based on array-comprehensive genome hybridization(aCGH), single nucleotide polymorphism array(SNP-array) or next generation sequencing(NGS), to be the most powerful technology. However, for whom this PGS technique is most suitable to achieve improved clinical outcome have not yet been identified by well defined, ITT based research with carefully selected control and adequate sample size.

The investigators research is to determine whether in vitro fertilization (IVF)/ intracytoplasmic sperm injection (ICSI) combined with SNP-array based pre-implantation comprehensive chromosome screening (CCS) will improve the clinical outcome of infertile female patients with recurrent spontaneous abortion history.

ELIGIBILITY:
Inclusion Criteria:

Women 18-48 years of age who are scheduled for IVF or ICSI with a history of recurrent spontaneous abortion (continous miscarriage occurred earlier than 20 weeks of gestation for equal or greater than 2 times) in our IVF institute while meeting the following criteria:

1. regular menstrual cycles and normal level of E2, P, FSH, LH, T, RPL in the early follicular phase;
2. no history of hormone medicine application in the last 3 months;
3. no history of poison contact;
4. normal uterine and adnexal ultrasonography;
5. TORCH(-), chlamydia(-), mycoplasma(-), normal leucorrhoea routine, anti-phospholipid antibody (-), antinuclear antibody(-);
6. for the couple, no blood type incompatibility or ABO antibody IgG≤1：64 and normal blood chromosome analysis.

Exclusion Criteria:

1. hydrosalpinx without operation; endometriosis; polycystic ovary syndrome; adenomyosis; uterine leiomyomata(submucous myoma or non-submucous myoma which size was exceed 4cm and/or with the compressed endometrium);uterine cavity lesions(such as uterine malformation, intrauterine adhesions, the septate uterus, endometritis etc);
2. the former abortion is because of luteal phase defect without treatment;
3. thyroid dysfunction or increased CA125 level;
4. acute inflammation of genitourinary system or STD carriers;
5. unable to comply with the study procedures.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 12 weeks after embryo transfer for the patient
  Ongoing pregnancy is defined as a viable intrauterine pregnancy after 12 weeks of embryo transfer.
  Ongoing pregnancy rate per treatment cycle will also be calculated on intend-to-treat(ITT) basis.

SECONDARY OUTCOMES:
Implantation of transferred embryo | 2 weeks after embryo transfer for the patient
  Implantation rate per embryo transferred will also be calculated.
Clinical pregnancy | 4 weeks after embryo transfer for the patient
  Clinical pregnancy is defined as the presence of a gestational sac confirmed by transvaginal ultrasound examination.
  Clinical pregnancy rate per treatment cycle will also be calculated based on ITT.
Time to pregnancy | from the date of the first time entering oocyte retrieval cycle until the embryo transfer day of a later assured ongoing pregnancy, accessed up to 24 months during the whole research period
  Time to pregnancy is defined as from the first time entering oocyte retrieval cycle to the embryo transfer day of a later assured ongoing pregnancy, which is up to 24 months within the study period. If the patient fails obtain ongoing pregnancy during the study period, the "time to pregnancy" will not be recorded for the specific patient or be calculated for the "average time to pregnancy" for the arm.
Pregnancy outcome | up to 42 days of a live birth
  abortion, live birth, multiple births, birth defect, preterm delivery, small-for-gestational age, still birth, maternal complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, MD, Study Director — Shanghai Jiai Genetics & IVF Institute; YILUN SUI, MD, Principal Investigator — Shanghai Jiai Genetics & IVF Institute
Locations (1):
- Shanghai Jiai Genetics & IVF Institute, Shanghai, China

REFERENCES:
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291